CLINICAL TRIAL: NCT05122936
Title: The Observation Study on Obesity Cohort Undergoing XRXPY-based Obesity Wellness Intervention
Brief Title: Observation on Obesity Undergoing XOWI
Status: Enrolling by invitation | Type: Observational
Sponsor: Feng Tao (Other)
Responsible Party: Sponsor-Investigator, Feng Tao, Director, Department of Endocrinology, Shanghai Municipal Hospital of Traditional Chinese Medicine
Organization: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Other Study IDs: SHMHTCM
Record Dates: First submitted 2021-10-24; First posted 2021-11-17 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Traditional Chinese Medicine
Keywords: Obesity; Traditional Chinese medicine; SRXPY-based Obesity Wellness Intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, feces, et al
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- XOWI Group: Obesity Cohort undergoing XRXPY-based Obesity Wellness Intervention
  Interventions: Combination Product: XRXPY-based Obesity Wellness Intervention(SOWI)

INTERVENTIONS:
Combination Product: XRXPY-based Obesity Wellness Intervention(SOWI) — It is an integrated obesity wellness intervention, composing of lifestyle invention and Chinese herbal therapy (XRXP granule, twice daily, oral administration). XRXPY is made in accordance with standard procedures. Participants will be instructed by TCM practitioner and educated by nutritionist. They will perform diet self-report by WeChat, recording daytime physical active steps and all-day sleeping time by electric bracelet. All the participants will be followed every 2-4 weeks by means of out-patient clinic, phone call or WeChat.

SUMMARY:
Obesity becomes a worldwide chronic health problem, including China. Meta-analyses showed in recent years anti-obesity effects of Chinese herbal therapy (CHT) in overweight and obese patients. However, there are still few observational studies on its effect in patients undergoing CHT more than 6 months, or on its safety. This is a mono-centric, prospective study conducted at Shanghai Municipal Hospital of Traditional Chinese Medicine. Patients with body mass index ≥ 28 Kg/m2 and chartered by heat-dampness is consecutively recruited. All the patients will undergo an integrated SRXPY-based Obesity Wellness Intervention (lifestyle invention + XRXP granule). Patients will be instructed by Traditional Chinese Medicine(TCM) practitioner and nutritionist. They will be investigated every 3 months, until 2 years after enrollment. The study will test anti-obesity effect and safety of the integrated obesity wellness intervention, and test changes of appetite, health-related quality of life, bio markers as well.

DETAILED DESCRIPTION:
Obesity is a worldwide problem to public health, with a prevalence rate of 12.4% according to recent studies. It is associated with a series of chronic non-communicable diseases, including type 2 diabetes, cardiovascular diseases, non-alcoholic fatty liver, polycystic ovary syndrome, cancer, and so on. Many publications reported Chinese herbal therapy as an effective anti- obesity management. However, there are still few observational studies on its effect in patients undergoing Chinese herbal therapy more than 6 months, or on its safety.

This is a mono-centric, prospective study conducted at Shanghai Municipal Hospital of Traditional Chinese Medicine. Patients with body mass index ≥ 28 Kg/m2 will be consecutively recruited in out-patient clinic of the department of endocrinology or nutrition. Another important including criteria is that each subject is supposed to be chartered by heat-dampness pattern in TCM. Patients will undergo an integrated SRXPY-based obesity wellness intervention(SOWI). They will report weekly diet, daytime physical activities and sleeping time, by means of WeChat and Electrical bracelet. Meanwhile, TCM practitioner and nutritionist will be involved in helping them.

The integrated obesity wellness intervention is based on lifestyle invention and XRXP granule. XRXP granule is composed of several herbs, such as Huang Qin (Baical Skullcap Root), Zi Cao (Root of Sinkiang Arnebia), Hu Zhang (Rhizoma Polygoni cuspidata), Cang Shu (Atractylodis Rhizoma), He Ye (Lotus Leaf), etc. Some components have been found, which can ameliorate serum concentrations of glucagon-like peptide-1 by stimulating gut taste receptors in db/db mice. Also, XRXP granule showed anti-obesity effects (reduction of body weight, body mass index and waist circumstance) in a 12-week pilot study on obese patients.

In this observational study, patients will be investigated every 3 months, until 2 years after enrollment. We will not only test the effect and safety, but test changes of appetite, health- related quality of life, bio markers as well.

ELIGIBILITY:
Inclusion Criteria:

·age ranged from 16-70 years old body mas index over 28kg/m2

Exclusion Criteria:

* secondary cause of obesity such as hypothalamic obesity, cushing syndrome, and hypophysis dysfunction, etc.
* pregnancy or lactation
* significant dysfunction of heart, liver, kidney and systemic organs (NYHA Class III or IV; alanine aminotransferase(ALT) and / or aspartate aminotransferase(AST) ≥ 5 times the normal upper limit; glomerular filtration rate< 60(ml/min) or with malignant tumor
* body weight fluctuated by more than 5 kg in the last 3 months with drug abuse or alcohol addiction
* with serious mental and neurological disorders
* blood pressure ≥ 180/110 mmHg, or malignant hypertension
* organic and systemic diseases intolerant of herb

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 Patients from the outpatient clinic of Shanghai Municipal Hospital of TCM will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Change in Body Weight | 2021-2027
  Measuring body weight at the required time point
Percentage of Participants who Achieve ≥5% Body Weight Reduction | 2021-2027
  Measuring body weight at the required time point

SECONDARY OUTCOMES:
Percentage of participants who achieve ≥10% body weight reduction | 2021-2027
  Measuring body weight at the required time point
Percentage of participants who achieve ≥15% body weight reduction | 2021-2027
  Measuring body weight at the required time point
Change in waist circumference | 2021-2027
  Measuring waist circumference at the required time point
Change in glycosylated hemoglobin A-1c(Hba1c) | 2021-2027
  Measuring Hba1c at the required time point
Change in fasting blood glucose | 2021-2027
  Measuring fasting blood glucose at the required time point
Change in Three-Factor eating questionnaire(TFEQ-R21) | 2021-2027
  Investigating TFEQ-R21 at the required time point
Change in food craving questionnaire-trait(FCQ-T) | 2021-2027
  Investigating FCQ-T at the required time point
Change in Impact of weight quality of life-lite(IWQOL-Lite) | 2021-2027
  Investigating IWQOL-Lite at the required time point，higher scores indicate better quality of life on the IWQOL-Lite(0-100).
Change in the medical outcomes study item short from health survey-short from(SF-36) | 2021-2027
  Investigating SF-36 at the required time point，higher scores indicate better quality of life on the SF-36(0-100).
Change in cholecystokinin(CCK) | 2021-2027
  Measuring CCK in serum at the required time point
Change in bile acid | 2021-2027
  Measuring bile acid in serum and feces at the required time point
Change in peptide YY(PYY) | 2021-2027
  Measuring PYY in serum at the required time point
Change in ghrelin(GHRL) | 2021-2027
  Measuring GHRL in serum at the required time point

CONTACTS AND LOCATIONS:
Overall Officials: Feng Tao, Study Director — Shanghai Municipal Hospital of Traditional Chinese Medicine
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data materials will publish articles